CLINICAL TRIAL: NCT07020039
Title: Comparing Photon Counting Computed Tomography With Invasive Coronary Angiography and Intravascular Ultrasound in Detecting Cardiac Allograft Vasculopathy
Brief Title: Comparing PCCT With ICA and IVUS in Detecting Cardiac Allograft Vasculopathy
Acronym: CAVIAR
Status: Not yet recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Kristjan Karason, MD, PhD, Sahlgrenska University Hospital
Other Study IDs: CAVIAR 2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Heart transplantation; Cardiac allograft vasculopathy; photon counting computed tomography; Invasive coronary angiography; Intravascular ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — Proteomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In traditional coronary artery disease, patients often experience symptoms such as angina. However, heart transplant patients lack nerve connections in the transplanted heart and therefore usually do not notice any symptoms. For this reason, routine examinations are performed using traditional coronary angiography at one, three, and six years after transplantation, sometimes with the addition of coronary ultrasound.

A new technique, photon-counting computed tomography, has now been developed and may potentially replace both traditional coronary angiography and intravascular ultrasound. In this study, we aim to investigate how well this method works in diagnosing coronary artery changes compared to the established methods.

DETAILED DESCRIPTION:
Cardiac allograft vasculopathy (CAV) is a major cause of graft failure and mortality in heart transplant recipients. Unlike traditional atherosclerosis, CAV is characterized by diffuse intimal hyperplasia and concentric narrowing of coronary arteries, affecting both epicardial vessels and the microvasculature. The cause is largely unknown, although it is believed that both immunologic and non-immunologic factors could be at play. CAV is frequently asymptomatic due to denervation of the transplanted heart, underscoring the importance of routine surveillance to enable early and accurate detection. Such monitoring is essential to optimize post-transplant outcomes.

Invasive coronary angiography (ICA) is the gold standard for diagnosing CAV, while intravascular ultrasound (IVUS) can be considered as the gold standard for the assessment of intimal thickening and plaque burden. Photon-counting computed tomography (PCCT) represents a novel, non-invasive imaging modality with superior spatial resolution and tissue contrast compared to conventional CT systems.

A systematic comparison of PCCT with ICA and IVUS for detecting CAV has not yet been performed. This study aims to assess the diagnostic accuracy, clinical relevance, and cost-effectiveness of PCCT in comparison to ICA and IVUS. By evaluating the advantages and limitations of non-invasive versus invasive modalities, the study seeks to define the optimal surveillance strategy for CAV, ultimately guiding the management of heart transplant recipients and improving long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult heart transplant recipients.
* Clinically stable and scheduled for routine ICA.
* Ability to provide informed consent

Exclusion Criteria:

* Contrast allergy
* Renal insufficiency with eGFR < 30 ml/min/m2
* Other contraindications for PCCT, ICA, or IVUS
* Acute cardiac events within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult heart transplant recipients scheduled for routine coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of PCCT compared to ICA in detecting CAV | 2 days
  Non-invasive investigation compared to invasive procedures
Level of agreement between PCCT and ICA in grading CAV severity | 2 days
  Non-invasive investigation compared with invasive procedures

SECONDARY OUTCOMES:
Correlation between PCCT and IVUS in quantifying lumen area, wall thickness, and plaque burden. | 2 days
  PCCT compared with IVUS
Radiation dose exposure using PCCT contra ICA/IVUS. | 2 days
  Radiation dose compared between PCCT and ICA/IVUS
Cost-effectiveness of PCCT versus ICA/IVUS | 2 days
  The cost of PCCT verus ICA/IVUS
Patient comfort and procedural time differences with PCCT versus IVA/IVUS | 2 days
  Comparing patient comfort during PCCT and ICA/IVUS, respectively

OTHER OUTCOMES:
Relationship between CAV and periarterial fat density as well as myocardial fibrosis | 1 day
  To see whether periarterial fat density and myocardial fibrosis are related to CAV

CONTACTS AND LOCATIONS:
Overall Officials: Kristjan Karason, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Transplant Institute, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 1 2028
Access Criteria: Reasonable request
URL: http://sahlgrenska.se

REFERENCES:
- [Background] Pober JS, Chih S, Kobashigawa J, Madsen JC, Tellides G. Cardiac allograft vasculopathy: current review and future research directions. Cardiovasc Res. 2021 Nov 22;117(13):2624-2638. doi: 10.1093/cvr/cvab259. PMID 34343276
- [Background] Velleca A, Shullo MA, Dhital K, Azeka E, Colvin M, DePasquale E, Farrero M, Garcia-Guereta L, Jamero G, Khush K, Lavee J, Pouch S, Patel J, Michaud CJ, Shullo MA, Schubert S, Angelini A, Carlos L, Mirabet S, Patel J, Pham M, Urschel S, Kim KH, Miyamoto S, Chih S, Daly K, Grossi P, Jennings DL, Kim IC, Lim HS, Miller T, Potena L, Velleca A, Eisen H, Bellumkonda L, Danziger-Isakov L, Dobbels F, Harkess M, Kim D, Lyster H, Peled Y, Reinhardt Z. The International Society for Heart and Lung Transplantation (ISHLT) guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2023 May;42(5):e1-e141. doi: 10.1016/j.healun.2022.10.015. Epub 2022 Dec 20. No abstract available. PMID 37080658
- [Background] Tavakol M, Ashraf S, Brener SJ. Risks and complications of coronary angiography: a comprehensive review. Glob J Health Sci. 2012 Jan 1;4(1):65-93. doi: 10.5539/gjhs.v4n1p65. PMID 22980117
- [Background] Sharma A, Cerdas MG, Reza-Soltani S, Rustagi V, Guntipalli M, Rojas Torres DS, Bhandari M, Kandel S, Teja Rayaprolu D, Hussain M. A Review of Photon-Counting Computed Tomography (PCCT) in the Diagnosis of Cardiovascular Diseases. Cureus. 2024 Nov 6;16(11):e73119. doi: 10.7759/cureus.73119. eCollection 2024 Nov. PMID 39650912